CLINICAL TRIAL: NCT00637702
Title: A Study of ARRY-334543 in Patients With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Array Biopharma, now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Organization: Array BioPharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARRAY-543-103
Record Dates: First submitted 2008-03-12; First posted 2008-03-18 (Estimated); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Advanced Cancer
MeSH Terms: interventions — ARRY-334543

ARMS (1):
- ARRY-334543 (Experimental)
  Interventions: Drug: ARRY-334543, EGFR/ErbB2 inhibitor; oral

INTERVENTIONS:
Drug: ARRY-334543, EGFR/ErbB2 inhibitor; oral — single dose and multiple dose, escalating

SUMMARY:
This is a Phase 1 study during which patients with advanced solid tumors will receive a new formulation of investigational study drug ARRY-334543. Patients will receive increasing doses of study drug in order to achieve the highest dose possible that will not cause unacceptable side effects. The patients will be followed to see what side effects and effectiveness the study drug has, if any, in treating the cancer. In addition, the effect of food on the new formulation will be evaluated. Approximately 24 patients from Canada will be enrolled in this study (Active, not recruiting).

ELIGIBILITY:
Key Inclusion Criteria:

* Histological or cytological evidence of malignancy.
* Patients with advanced solid tumors who are no longer candidates for standard therapy, have no standard therapy available, or choose not to pursue standard therapy.
* Cardiac ejection fraction ≥ 50% by echocardiogram (ECHO) or multiple gated acquisition (MUGA).
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0, 1 or 2.
* Additional criteria exist.

Key Exclusion Criteria:

* Uncontrolled brain metastases (if a patient has brain metastases and is on steroids, the steroid dose must be stable for at least 30 days).
* Use of an investigational medication or device within 30 days prior to first dose of study drug.
* Major surgery within 30 days prior to first dose of study drug.
* Radiotherapy or chemotherapy within 28 days prior to first dose of study drug (not including palliative radiotherapy at focal sites).
* Active, uncontrolled infection requiring systemic antibiotic therapy or other serious underlying medical condition which would impair the ability of the patient to receive protocol treatment.
* Pregnancy or lactation.
* Known positive serology for the human immunodeficiency virus (HIV), 'active' hepatitis B and/or hepatitis C.
* Additional criteria exist.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2008-02; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Characterize the safety profile of the new formulation of study drug in terms of adverse events, clinical laboratory tests and electrocardiograms. | Duration of study
Establish the maximum tolerated dose (MTD) of the new formulation of study drug. | Duration of study
Characterize the pharmacokinetics (PK) of the new formulation of study drug (in terms of plasma concentrations) when administered in a fed versus fasted state. | Day 1 and Day 8
Assess the exposure of the new formulation of study drug in terms of plasma concentrations. | Duration of study

SECONDARY OUTCOMES:
Assess the efficacy of the new formulation of study drug in terms of tumor dimension assessment. | Duration of study

CONTACTS AND LOCATIONS:
Overall Officials: Pizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- Canada (2):
  - Juravinski Cancer Center at Hamilton Heath Sciences, Hamilton, Ontario
  - Ottawa Hospital Cancer Centre, Ottawa, Ontario